CLINICAL TRIAL: NCT00479596
Title: Safety and Efficacy Study of Intradetrusor Injections of Botox® for the Treatment of Urinary Incontinence Secondary to Benign Prostatic Obstruction (BTX0621)
Brief Title: This is a Prospective, Randomized, Double-Blind Study Comparing Intravesical Injection of Botox® to Placebo.
Acronym: BTX0621
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Urological Sciences Research Foundation (Other)
Collaborators: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTX0621
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-01

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; OAB; Refractory OAB; Botox; Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botox

SUMMARY:
The current study will investigate the comparative efficacy, safety and patient satisfaction of intradetrusor injections BOTOX® injections (200U) versus placebo (saline) injections in the treatment of OAB secondary to benign prostatic obstruction (BPO).

DETAILED DESCRIPTION:
Overactive bladder is a common problem that follows chronic prostatic bladder outlet obstruction and is part of the benign prostatic hyperplasia syndrome (BPH) in men. Unfortunately, it does not often resolve after treatment (TURP, etc) of the obstruction from enlarged prostate gland. Patients with obstructive BPH typically commence treatment with alpha-blockers or anticholinergic agents; the former being used to treat enlarged prostate medically, and the latter to treat overactive bladder symptoms. However, as mentioned, anticholinergics cause many intolerable side effects leading to discontinuation in many patients. Furthermore this class of drug is still considered a relative contraindication in this population by some clinicians. Therefore other modalities need to be studied in these men.

Based on numerous studies in overactive bladder (OAB), we hypothesize that these patients will experience significant improvement (particularly if their symptoms of urgency and frequency) without significant side effects from intradetrusor injections of BOTOX® even though they have were refractory to systemic anticholinergics.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 40 and 90 years of age.
2. Clinical signs and symptoms of frequency and urgency
3. Urodynamic history consistent with OAB that developed in conjunction with Benign Prostate Obstruction and that persists for at least 3 months post TURP or PVP, or other obstruction relieving procedure.
4. OAB inadequately controlled with anticholinergic medications
5. Qmax >12mL/s with a voided volume of >125mL.
6. IPSS >12, with IPSS QoL >3 at study Visit 1.
7. Willing to use clean intermittent catheterization (CIC) to empty the bladder or is willing to have an indwelling catheter, if necessary following study treatment.

Exclusion Criteria:

1. Known history of interstitial cystitis, uninvestigated hematuria, bladder outlet obstruction due to vesical neck contracture, mullerian duct cysts, urethral obstruction due to stricture/valves/sclerosis of urethral tumor, radiation cystitis, genitourinary tuberculosis, bladder calculi, or detrusor-sphincter dyssynergia.
2. Current indwelling catheter, or removal of chronic catheter <1 month prior to study entry.
3. Non-compliance with wash-out periods for prohibited medications/therapies
4. Evidence of Urinary Tract Infection according to local standard of care.
5. History of prostate cancer.
6. Serum PSA of >10ng/mL. [NOTE: Subjects with serum PSA concentrations >4 and <10 must have prostate cancer excluded according to the local standard of care.]
7. 24 hour total volume voided >3000 mL of urine
8. Medical condition that may increase their risk of exposure to botulinum toxin including diagnosed Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis or any other disease that might interfere with neuromuscular function.
9. Allergy or sensitivity to any component of BOTOX®

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of BOTOX to placebo (saline) in the treatment of OAB secondary to BPO. | 6 months post injection

SECONDARY OUTCOMES:
Patient satisfaction to intradetrussor injection of Botox versus placebo. | 6 months post injection

CONTACTS AND LOCATIONS:
Overall Officials: Leonard S Marks, M.D., Principal Investigator — Urological Sciences Research Foundation
Locations (1):
- Urological Sciences Research Foundation, Culver City, California, United States

REFERENCES:
- See also: Related Info — http://www.usrf.org